CLINICAL TRIAL: NCT02442024
Title: Metabolic Effects of the Manipulation of Nutrient Sequence in the Main Meals in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Andrea Natali, Professor, Azienda Ospedaliero, Universitaria Pisana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPPO
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; diet; nutrient sensing
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified diet (Experimental): This group will follow a modified diet over a period of two months.
  Interventions: Behavioral: Modified Diet
- Standard diet (Active Comparator): This group will follow a standardized diet over a period of two months.
  Interventions: Behavioral: Standard Diet

INTERVENTIONS:
Behavioral: Modified Diet — Two months of a diet in which the ingestion of protein and lipid precedes that of carbohydrates.
  Arms: Modified diet
Behavioral: Standard Diet — Two months of a diet in which the ingestion of protein and lipid follows that of carbohydrates.
  Arms: Standard diet

SUMMARY:
The investigators aimed at evaluating the metabolic effects of the inversion of the typical Italian sequence of food ingestion at the main meals in type 2 diabetic patients.

DETAILED DESCRIPTION:
An intervention group follows a modified diet over a period of two months in which the ingestion of protein and lipid happens before that of carbohydrates. A control group follows a standardized diet in which the ingestion of carbohydrates happens before that of protein and lipid. Both diets contain a reduced intake of high-glycemic index meals, saturated fatty acids, trans fatty acids and alcohol.

On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet) we measure clinical and metabolic parameters (weight, waist and hip circumferences, glucose, glycated hemoglobin, fructosamine, lipid profile) to compare the effects of the two diets.

ELIGIBILITY:
Inclusion Criteria:

* Well-controlled type 2 diabetes
* HbA1c 48-58 mmol/mol (6.5-7.5%)
* Treatment with metformin or diet only
* BMI: < 35 kg/m^2

Exclusion Criteria:

* Autoimmune diseases, neoplasia, heart, kidney, liver or respiratory failure
* Pregnancy
* Bariatric surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline fructosamine after 1 and 2 months of diet | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Fructosamine will be measured.

SECONDARY OUTCOMES:
Change from baseline fasting plasma glucose after 1 and 2 months of diet | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Fasting plasma glucose will be measured.
Change from baseline glycated hemoglobin after 1 and 2 months of diet | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Glycated hemoglobin will be measured.
Change from baseline weight after 1 and 2 months of diet adipose tissue location | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Waist circumference and hip circumference will be measured.
Change from baseline adipose tissue location after 1 and 2 months of diet | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Weight, waist circumference and hip circumference will be measured.
Change from baseline lipid profile after 1 and 2 months of diet | On four days separated by one month each other (two before the beginning of the diet and two after 1 month and 2 months of diet)
  Lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natali, Professor, Study Chair — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy